CLINICAL TRIAL: NCT03392935
Title: Efficacy of 1540 Nanometer Erbium Glass Laser to Improve Benign Dermatofibromas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_101842
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Results first posted 2021-06-23 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2021-06

CONDITIONS: Dermatofibroma of Skin

STUDY DESIGN:
Intervention Model Description: All subjects will have their dermatofibromas treated with the laser at week 0, and week 4. Blinded outcome assessors will rate photos (pre-treatment and follow-up visit 1) to determine efficacy.
Masking Description: Outcome assessors are masked and will not know which photos are pre-treatment or follow-up visit 1, however, they do know that all subjects received treatment at some point. They will rate the dermatofibromas to determine efficacy. However, there is only one arm of this study. All patients are receiving the same treatment. Outcomes assessors are the only masked roles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All Subjects (Experimental): All subjects will be treated with the laser at week 0 and week 4. Only assessors will be blinded and rate the dermatofibromas in photographs, they will not know which photos were taken pre-treatment vs. post-treatment to determine efficacy.
  Interventions: Device: 1540 nanometer Erbium glass laser

INTERVENTIONS:
Device: 1540 nanometer Erbium glass laser — Subjects will receive laser treatment by dermatologist at week 0 and week 4.

SUMMARY:
This study is to find a more effective treatment for itchy, painful or unsightly dermatofibromas, that will improve symptoms of itch and/or pain and/or improve the appearance of dermatofibromas. This is an open-label study where subjects will receive a laser treatment at week 0, and week 4, and then 2 additional follow-up visits. Photographs will be taken at each visit and rated by blinded reviewers after the study to determine efficacy.

DETAILED DESCRIPTION:
The main objective of this study is to find a more effective treatment for itchy, painful or unsightly dermatofibromas, that will improve symptoms of itch and/or pain and/or improve the appearance of dermatofibromas. A secondary objective of this study is to better understand the 1540 nanometer Erbium glass laser and its impact on the skin.

This is an open-label study where subjects will receive a laser treatment at week 0, and week 4, and then have 2 additional follow-up visits (no laser treatment at these visits). Photographs will be taken at each visit and photographs from pre-treatment and follow-up 1 (week 8) will rated by blinded reviewers after the study to determine efficacy.

ELIGIBILITY:
Inclusion Criteria:

* female or male, age 18-65, have at least one dermatofibroma of the skin, on the trunk or extremities, diagnosed by dermatologist, dermatofibroma is either itchy, painful or unattractive to the patient.

Exclusion Criteria:

* previous treatment to the dermatofibroma(s), pregnant or nursing women, diabetic, smoker, psoriasis, lupus or other autoimmune diseases, patient with a clear history of keloids or poor wound healing. This study will exclude dermatofibroma lesions on the face and genitals.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Stolman, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- University of Utah Dermatology, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: lesions
Period: Overall Study
Arm/Group | All Subjects
Started | 37; 46 lesions
Completed | 35; 44 lesions
Not Completed | 2; 2 lesions

BASELINE CHARACTERISTICS:
Units Other Than Participants: Lesions
Arm/Group | All Subjects
Number analyzed (Participants) | 37
Number analyzed (Lesions) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Modified Patient and Observer Scar Assessment Scale Color Component Comparing Change From Baseline to Week 12.
Description: Patient reported assessment scale of pain, itch, color, and texture. Each element (pain, itch, color, and texture) is graded on a 1-10 scale.
  The lowest score is '1', which corresponds to the situation of normal skin/no symptoms (i.e. not different in color, not different in texture, no itching, no pain). Score 10 equals the largest difference from normal skin (i.e. severely painful, severely itchy, vert different color, very different texture).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: lesions
Arm/Group | All Subjects
Number analyzed (Participants) | 35
Number analyzed (lesions) | 44
score on a scale | -2.33 (2.33)

2. Secondary Outcome: Modified Patient and Observer Scar Assessment Scale Itch Component Comparing Change From Baseline to Week 12.
Description: as for outcome 1
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: lesion
Arm/Group | All Subjects
Number analyzed (Participants) | 35
Number analyzed (lesion) | 44
score on a scale | -0.25 (1.03)

3. Secondary Outcome: Modified Patient and Observer Scar Assessment Scale Texture Component Comparing Change From Baseline to Week 12.
Description: as for outcome 1
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: lesions
Arm/Group | All Subjects
Number analyzed (Participants) | 35
Number analyzed (lesions) | 44
score on a scale | -2.92 (2.89)

4. Secondary Outcome: Modified Patient and Observer Scar Assessment Scale Pain Component Comparing Change From Baseline to Week 12.
Description: as for outcome 1
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: lesions
Arm/Group | All Subjects
Number analyzed (Participants) | 35
Number analyzed (lesions) | 44
score on a scale | 0 (0.42)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to week 12.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 37/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=37)
Transient Erythema (Skin and subcutaneous tissue disorders) | 37 (87) — Transient expected redness at the site of laser applicaiton, resolving within 3 days of treatment without sequela. .
Transient Edema (Skin and subcutaneous tissue disorders) | 37 (87) — Transient expected swelling at site of laser application, resolving within 3 days of treatment without sequela.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT03392935/Prot_SAP_002.pdf
  • Informed Consent Form (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT03392935/ICF_001.pdf